CLINICAL TRIAL: NCT00938535
Title: Community Based Obesity Prevention Among Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2628; 1R01DK078798 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Obesity; Women's health; Minority health; Obesity prevention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obesity Prevention (Experimental)
  Interventions: Behavioral: Obesity Prevention
- Usual Care (No Intervention): This arm includes usual care.

INTERVENTIONS:
Behavioral: Obesity Prevention — This arm includes an action plan, tailored print materials, telephone support calls, interactive self-monitoring, and a 12-month YMCA membership for the participant.
  Arms: Obesity Prevention

SUMMARY:
This study will evaluate the efficacy of a behavioral intervention, designed to prevent weight gain among overweight and low obese (25-34.9 kg/m2) Black women (aged 25-44), compared to usual care.

DETAILED DESCRIPTION:
Obesity prevention among Black women is a major public health priority; presently, nearly 54% of the adult Black female population is obese. To date, most intervention attention has been focused on weight reduction among the overweight and obese. However, both conditions are notoriously recalcitrant to treatment, particularly among Blacks. We posit that obesity prevention might represent a particularly effective intervention strategy for overweight Black women. Most studies have shown that Black women have a greater social acceptance of overweight, less body weight dissatisfaction, and higher ideal body weights, compared to Whites. Furthermore, numerous studies have shown that obesity is less lethal and causes fewer co-morbidities among Black vs. White women, suggesting that maintaining overweight may be an appropriate public health goal for Black women. We posit that an intervention approach that emphasizes maintaining overweight, while preventing the transition to obesity will resonate among the target population. Very few obesity prevention RCTs appear in the published literature and, to our knowledge, none have been conducted solely among Black women.

We propose to randomize overweight, Black women (n=184) to either usual care (UC) or an obesity prevention (OP) intervention condition. The OP condition is comprised of several intervention components that will be delivered over 12 months; each participant will receive a tailored action plan, tailored print materials, monthly coaching calls, and weekly self-monitoring via an interactive voice response system. Assessments will be taken at baseline, 6, 12, and 18 months post baseline.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* Female
* Ages 25-44
* BMI between 25-34.9 kg/m2
* Patients with at least 1 visit in the previous 24 months to a participating Community Health Center

Exclusion Criteria:

* Not currently pregnant
* Not given birth within the past 12 months
* No history of myocardial infarction or stroke in last 2 years

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in BMI. We have set a target of BMI maintenance among those randomized to the intervention condition. | 6, 12 and 18 months post baseline

SECONDARY OUTCOMES:
Change in obesity risk behaviors | 6, 12 and 18 months post baseline
Measures of body composition | 6, 12 and 18 months post baseline
Psychosocial mediators | 6, 12 and 18 months post baseline
Obesity related biomarkers | 6, 12 and 18 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Result] Bennett GG, Foley P, Levine E, Whiteley J, Askew S, Steinberg DM, Batch B, Greaney ML, Miranda H, Wroth TH, Holder MG, Emmons KM, Puleo E. Behavioral treatment for weight gain prevention among black women in primary care practice: a randomized clinical trial. JAMA Intern Med. 2013 Oct 28;173(19):1770-7. doi: 10.1001/jamainternmed.2013.9263. PMID 23979005
- [Derived] Gallis JA, Kusibab K, Egger JR, Olsen MK, Askew S, Steinberg DM, Bennett G. Can Electronic Health Records Validly Estimate the Effects of Health System Interventions Aimed at Controlling Body Weight? Obesity (Silver Spring). 2020 Nov;28(11):2107-2115. doi: 10.1002/oby.22958. Epub 2020 Sep 27. PMID 32985131
- [Derived] Greaney ML, Askew S, Wallington SF, Foley PB, Quintiliani LM, Bennett GG. The effect of a weight gain prevention intervention on moderate-vigorous physical activity among black women: the Shape Program. Int J Behav Nutr Phys Act. 2017 Oct 16;14(1):139. doi: 10.1186/s12966-017-0596-6. PMID 29037247
- [Derived] Steinberg DM, Christy J, Batch BC, Askew S, Moore RH, Parker P, Bennett GG. Preventing Weight Gain Improves Sleep Quality Among Black Women: Results from a RCT. Ann Behav Med. 2017 Aug;51(4):555-566. doi: 10.1007/s12160-017-9879-z. PMID 28213632
- [Derived] Steinberg DM, Levine EL, Lane I, Askew S, Foley PB, Puleo E, Bennett GG. Adherence to self-monitoring via interactive voice response technology in an eHealth intervention targeting weight gain prevention among Black women: randomized controlled trial. J Med Internet Res. 2014 Apr 29;16(4):e114. doi: 10.2196/jmir.2996. PMID 24780934
- [Derived] Foley P, Levine E, Askew S, Puleo E, Whiteley J, Batch B, Heil D, Dix D, Lett V, Lanpher M, Miller J, Emmons K, Bennett G. Weight gain prevention among black women in the rural community health center setting: the Shape Program. BMC Public Health. 2012 Jun 15;12:305. doi: 10.1186/1471-2458-12-305. PMID 22537222